CLINICAL TRIAL: NCT02185547
Title: Effects and Consequences for Mother and Child From Treatment for Depression, A Prospective Randomized, Placebo- Controlled, Trial With Internet-based Cognitive Behavior Therapy and Sertraline or Placebo for Moderate Depression in Pregnancy
Brief Title: Effects and Consequences for Mother and Child From Treatment for Depression
Acronym: MAGDALENA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties in recruiting participants.
Sponsor: Katarina Wide (Other)
Responsible Party: Sponsor-Investigator, Katarina Wide, M.D associated professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KWMP001
Record Dates: First submitted 2014-07-06; First posted 2014-07-09 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Pregnancy; Moderate Depression
Keywords: women
MeSH Terms: interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICBT in combination with sertraline treatment (Experimental): Internet cognitive behavioral therapy in combination with sertraline treatment
  Interventions: Drug: Zoloft; Behavioral: ICBT
- ICBT (Active Comparator): Only Internet cognitive behavioral treatment, no additional depression treatment
  Interventions: Behavioral: ICBT

INTERVENTIONS:
Drug: Zoloft — Sertraline treatment 25 mg
  Arms: ICBT in combination with sertraline treatment
Behavioral: ICBT — Internet behavioral cognitive therapy only

SUMMARY:
This study targets women with moderate depression during pregnancy. We aim to investigate the direct effect of the newborn child and the long term consequences on the cognitive developement on children who´s mother has been treated with CBT alone or in combination with antidepressants.

DETAILED DESCRIPTION:
The primary objective is to study the direct neonatal effects and the long-term consequences on cognitive development in children prenatal exposed to maternal sertraline treatment compared to exposure to maternal depression treated with only ICBT.

ELIGIBILITY:
Inclusion Criteria:

1. Female > 18 years old
2. Pregnant, gestational week 9-21.
3. Verified moderate depression according to SCID-I with or without concomitant anxiety disorder.
4. Signed informed consent
5. Able to understand the Swedish language orally and in written and able to use the internet for the ICBT, including having succeded in filling out online questionnaires
6. Are willing to participate to all study visits
7. Plans to give birth at the Department of Obstetrics at Karolinska University Hospital, Huddinge or at additional study site such as Norrland University Hospital (NUS), Umeå

Exclusion Criteria:

* 1. Known drug or alcohol abuse 2. Serious psychiatric disorder such as psychosis, bipolar disorder, severe personality disorder, ADHD/ADD, autism or mental retardation) and severe melancholic or psychotic depression.

  3. Known idiosyncrasy to Zoloft or allergy to one of the Zoloft excipients 4. Ongoing medication with SSRI, SNRI, TCA, mood-stabilizers, antiepileptic drugs ,psychotropic drugs, tramadol, propafenon, tolbutamid, flekainid, psychostimulants and atomoxetine, insulin or steroids 5. Any severe somatic disease that necessitate regular treatment with systemic steroids, severe heart and lung disease, kidney disease, liver disease, diabetes mellitus, or epilepsy with drug treatment.

  6. Women who either during screening or treatment on self-assessment forms (MADRS-S: 4 or more points on question about suicidal ideation (question 9)) report symptoms of severe suicidal thoughts or suicide plans will be contacted for structured suicide risk assessment by telephone (by experienced staff from the unit for internet psychiatry according to clinical routine). If judged necessary patients will be booked for psychiatric assessment by study nurse. If acute assessment or care is judged necessary, referral to psychiatric emergency departments will be made according to the same routine as in regular care.

Also women, who contact the study personal and report symptoms of suicidal thoughts or suicide plans will receive psychiatric assessment as specified above. Women who according to psychiatric assessment have a high suicidal risk will be excluded from the study. These women will be actively transferred into necessary psychiatric treatment as usual.

7. Other factors that are clinical significant and could jeopardize study results or its intention, as judged by study psychiatrist or study obstetrician

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-02-21 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Cognitive development | 2 years
  The differences in cognitive development at 2 years evaluated by the standard Bayley Scales of Infant and Toddler Development third edition (BSID-III)®.

SECONDARY OUTCOMES:
measure in MADRS_S | 12 weeks, 14 weeks and 30 weeks
  a) Add-on effect of sertraline measured in difference i) in self-report of depressive symptoms (MADRS-S),ii) in rate of remission from depression (measured by diagnostic psychiatric interview with MADRS at -12weeks, 14 weeks, and 30 weeks (= 3 months postpartum) of treatment
Stresshormone level | up to 3 months postpartum
  Effects on levels of S-hCG, cytokines,
Pharmacological assessment | 4, 14, 18 weeks
  Plasma sertraline concentrations.
Pharmacological assessment | 4, 14, 18 weeks
  Pharmacokinetic variations in the metabolism of sertraline. Assess activity of enzymes regulating the metabolism of sertralin.
Pharmacological assessment | 4, 14, 18 weeks
  Genetic variations in the metabolism of sertraline. Assess concentration of sertralin and markers for metabolism of sertralin on specific regions of sertralin pathways.
Pharmacological assessment | 4, 14, 18 weeks
  Effects on prolactin levels. Assess prolactin.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Wide K, Winbladh B, Kallen B. Major malformations in infants exposed to antiepileptic drugs in utero, with emphasis on carbamazepine and valproic acid: a nation-wide, population-based register study. Acta Paediatr. 2004 Feb;93(2):174-6. doi: 10.1080/08035250310021118. PMID 15046269
- [Background] Wide K, Winbladh B, Tomson T, Sars-Zimmer K, Berggren E. Psychomotor development and minor anomalies in children exposed to antiepileptic drugs in utero: a prospective population-based study. Dev Med Child Neurol. 2000 Feb;42(2):87-92. doi: 10.1017/s0012162200000177. PMID 10698324
- [Background] Pilo C, Wide K, Winbladh B. Pregnancy, delivery, and neonatal complications after treatment with antiepileptic drugs. Acta Obstet Gynecol Scand. 2006;85(6):643-6. doi: 10.1080/00016340600604625. PMID 16752253
- [Background] Wide K, Winbladh B, Tomson T, Kallen B. Body dimensions of infants exposed to antiepileptic drugs in utero: observations spanning 25 years. Epilepsia. 2000 Jul;41(7):854-61. doi: 10.1111/j.1528-1157.2000.tb00253.x. PMID 10897157
- [Background] Wide K, Henning E, Tomson T, Winbladh B. Psychomotor development in preschool children exposed to antiepileptic drugs in utero. Acta Paediatr. 2002;91(4):409-14. doi: 10.1080/080352502317371643. PMID 12061356
- [Background] Tomson T, Battino D, French J, Harden C, Holmes L, Morrow J, Robert-Gnansia E, Scheuerle A, Vajda F, Wide K, Gordon J. Antiepileptic drug exposure and major congenital malformations: the role of pregnancy registries. Epilepsy Behav. 2007 Nov;11(3):277-82. doi: 10.1016/j.yebeh.2007.08.015. PMID 17996635
- [Background] Fahnehjelm KT, Wide K, Ygge J, Hellstrom A, Tomson T, Winbladh B, Stromland K. Visual and ocular outcome in children after prenatal exposure to antiepileptic drugs. Acta Ophthalmol Scand. 1999 Oct;77(5):530-5. doi: 10.1034/j.1600-0420.1999.770509.x. PMID 10551294
- [Background] Forsberg L, Wide K, Kallen B. School performance at age 16 in children exposed to antiepileptic drugs in utero--a population-based study. Epilepsia. 2011 Feb;52(2):364-9. doi: 10.1111/j.1528-1167.2010.02778.x. Epub 2010 Nov 3. PMID 21054354
- [Derived] Heinonen E, Blennow M, Blomdahl-Wetterholm M, Hovstadius M, Nasiell J, Pohanka A, Gustafsson LL, Wide K. Sertraline concentrations in pregnant women are steady and the drug transfer to their infants is low. Eur J Clin Pharmacol. 2021 Sep;77(9):1323-1331. doi: 10.1007/s00228-021-03122-z. Epub 2021 Mar 22. PMID 33751155